CLINICAL TRIAL: NCT01257984
Title: A Multicenter, Open-label, Randomized, Controlled, Two-arm Study to Assess Compliance With Daily Tablet Intake of Women on Treatment With the Oral Contraceptive SH T00186D/BAY 86-5300 (0.02 mg Ethinyl Estradiol as Betadex Clathrate and 3 mg Drospirenone) in a Flexible Extended Regimen Supported by a Dispenser With a Reminder Function Over 12 Months
Brief Title: Study to Investigate Compliance With the Oral Contraceptive SH T00186D in a Flexible Extended Regimen Supported by a Dispenser With a Reminder Function
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14701; 2010-019902-17 (EudraCT Number)
Record Dates: First submitted 2010-12-09; First posted 2010-12-10 (Estimated); Last update posted 2014-10-28 (Estimated); Status verified 2014-10

CONDITIONS: Contraception

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: BAY86-5300
- Arm 2 (Experimental)
  Interventions: Drug: BAY86-5300

INTERVENTIONS:
Drug: BAY86-5300 — 0.02 mg EE as ß-CDC / 3 mg DRSP in a tablet form (1 tablet/day) for up to 120 days, followed by a 4-day tablet-free interval, administered with a dispenser supported by a reminder function
  Arms: Arm 1
Drug: BAY86-5300 — 0.02 mg EE as ß-CDC / 3 mg DRSP in a tablet form (1 tablet/day) for up to 120 days, followed by a 4-day tablet-free interval, administered with a dispenser without reminder support
  Arms: Arm 2

SUMMARY:
The objective of the study is to evaluate the effect of the dispenser's buzzer function on compliance with daily tablet intake of an ethinyl estradiol (EE) + drospirenone (DRSP) containing oral contraceptive (OC) in a flexible extended regimen when administered for approximately 12 months to healthy female volunteers who request contraception.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female volunteers between 18 and 35 years of age (smokers up to 30 years, inclusive) who request contraceptive protection

Exclusion Criteria:

* Pregnancy or lactation (less than 3 months since delivery, abortion, or lactation before start of treatment)
* Body mass index (BMI) >/= 30.0 kg/m2
* Presence or a history of venous or arterial thrombotic/thromboembolic events
* Repeated measurements of systolic blood pressure > 140 mmHg and/or diastolic blood pressure > 90 mmHg.
* Presence or history of liver tumors (benign or malignant), severe hepatic disease, jaundice and/or pruritus related to cholestasis, cholestatic jaundice associated with pregnancy or previous COC use
* Uncontrolled diabetes mellitus and/or diabetes mellitus with vascular involvement
* Severe dyslipoproteinemia
* Malignant or premalignant disease
* Uncontrolled thyroid disorder
* Chronic inflammatory bowel disease
* Severe renal insufficiency or acute renal failure
* History of migraine with focal neurologic symptoms
* Epilepsy

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 508 (Actual)
Dates: Start 2010-12; Primary Completion 2012-08 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Mean daily delay of tablet release, i.e. the time of tablet-release which will be compared to the reference tablet release time | 12 months

SECONDARY OUTCOMES:
Number of delayed and missed pills | 12 months
Bleeding pattern and cycle control parameters | 12 months
Length of the tablet break and the length of the bleeding episode preceding the tablet break | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (41):
- France (8):
  - Paris, Paris
  - Biarritz
  - Marly-le-Roi
  - Nancy
  - Olivet
  - Paris
  - Strasbourg
  - Toulouse
- Germany (9):
  - Heidelberg, Baden-Wurttemberg
  - Hamburg, Hamburg
  - Frankfurt am Main, Hesse
  - Wuppertal, North Rhine-Westphalia
  - Blankenburg, Saxony-Anhalt
  - Burg, Saxony-Anhalt
  - Magdeburg, Saxony-Anhalt
  - Gera, Thuringia
  - Kahla, Thuringia
- Italy (12):
  - Bologna
  - Brescia
  - Cagliari
  - Catania
  - Milan
  - Modena
  - Napoli
  - Palermo
  - Pavia
  - Pisa
  - Roma
  - Siena
- Spain (5):
  - Elda, Alicante
  - Barcelona, Barcelona
  - Córdoba, Córdoba
  - Boadilla del Monte, Madrid
  - Málaga, Málaga
- United Kingdom (7):
  - Chesterfield, Derbyshire
  - Nottingham, Nottinghamshire
  - Bath, Somerset
  - East Horsley, Surrey
  - Bradford-on-Avon, Wiltshire
  - Corsham, Wiltshire
  - Cardiff

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/